CLINICAL TRIAL: NCT00840970
Title: A Clinical Evaluation of the Steroid-Eluting Sinexus Intranasal Splint Used Following Functional Endoscopic Sinus Surgery (FESS) in Patients With Chronic Rhinosinusitis (CRS)
Brief Title: A Clinical Evaluation of the Sinexus Intranasal Splint Following Functional Endoscopic Sinus Surgery in Patients With Chronic Rhinosinusitis
Acronym: CONSENSUS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P500-0208
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Intervention Model Description: Intra-patient control where one ethmoid sinus was randomized to receive the intervention (treatment arm) while the contralateral ethmoid received the active comparator (control arm)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Efficacy Unilateral Control (Active Comparator): Non-coated splint placed unilaterally in the ethmoid sinus opening randomized to receive the active comparator following FESS (control arm)
  Interventions: Device: non-coated Intranasal Splint
- Efficacy Unilateral Treatment (Experimental): Drug-coated splint placed unilaterally in the ethmoid sinus opening randomized to receive the intervention following FESS (treatment arm)
  Interventions: Device: Sinexus Intranasal Splint
- Safety/PK Bilateral Treatment (Experimental): Drug-coated splints placed bilaterally in both ethmoid sinus openings following FESS
  Interventions: Device: Sinexus Intranasal Splint

INTERVENTIONS:
Device: non-coated Intranasal Splint — placement of non-coated intranasal splint following FESS
  Arms: Efficacy Unilateral Control
Device: Sinexus Intranasal Splint — placement of Sinexus Intranasal Splint placed following FESS
  Arms: Efficacy Unilateral Treatment; Safety/PK Bilateral Treatment

SUMMARY:
The purpose of this study is to assess the safety and performance of the Sinexus Intranasal Splint when used following Functional Endoscopic Sinus Surgery (FESS) in patients with Chronic Rhinosinusitis.

DETAILED DESCRIPTION:
This was a prospective, multi-center, double blind trial that enrolled patients in three groups as described below. Two groups (Pilot 15 mm and Efficacy 25 mm) used a randomized, double-blind, intra-patient control study design to assess performance of the drug-coated Splint (received in one ethmoid sinus) compared to the control Splint (received in the contralateral ethmoid). The other group of patients (Safety/PK 25 mm) received bilateral drug-coated Splints, and served as a pharmacokinetics (PK) study group.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient has a diagnosis of bilateral CRS defined as inflammation of the mucosa of the nose and paranasal sinuses of at least 12 consecutive weeks' duration.
* Patient has a clinical indication for and has consented to bilateral FESS.
* CRS diagnosis documented by CT scan within 60 days of the procedure.
* Patient has minimal total CT stage (Lund-Mackay method) of 6.
* Patient has bilateral disease defined as minimal CT stage per side of ≥3.

Exclusion Criteria:

* Oral-Steroid dependent COPD, asthma or other condition.
* Immune deficiency (IGG subclass deficiency or IGA deficiency).
* Symptomatic coronary artery disease.
* Patient undergoing chemotherapy treatment.
* Morbid obesity (BMI > 40) or a BMI that, in the opinion of the physician, would compromise health and participation in the study.
* Evidence of active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanier, MD, Principal Investigator — Central California Ear, Nose, Throat
Locations (1):
- Central California Ear, Nose, Throat, Fresno, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: ethmoid sinuses
Groups:
- Pilot 15 mm: First 7 patients (n=7) in the Pilot Phase received 15 mm length splint. This phase used a randomized intra-patient design wherein following FESS a non-coated splint was placed unilaterally in the ethmoid sinus opening randomized to receive the active comparator (control arm), and the drug-coated Sinexus Splint (15mm length, 220 ug mometasone furoate [MF]) was placed contralaterally in the ethmoid sinus opening randomized to receive the intervention (treatment arm). 15 mm length splint was not commercialized.
- Efficacy 25 mm: Efficacy group received the 25mm splint in the Pilot (n=13) and Pivotal Phases (n=25).
  Both phases used a randomized intra-patient design wherein following FESS a non-coated splint was placed unilaterally in the ethmoid sinus opening randomized to receive the active comparator (control arm), and the drug-coated Sinexus Splint (25 mm length, 370 ug MF) was placed contralaterally in the ethmoid sinus opening randomized to receive the intervention (treatment arm).
- Safety/PK 25 mm: Safety/PK group (n=5) used a non-randomized design wherein following FESS a drug-coated splints (25 mm length with 370 ug MF) were placed bilaterally in both ethmoid sinus openings.
Period: Overall Study
Arm/Group | Pilot 15 mm | Efficacy 25 mm | Safety/PK 25 mm
Started | 7; 14 ethmoid sinuses | 38; 76 ethmoid sinuses | 5; 10 ethmoid sinuses
Completed | 7; 14 ethmoid sinuses | 38; 76 ethmoid sinuses | 4; 8 ethmoid sinuses
Not Completed | 0; 0 ethmoid sinuses | 0; 0 ethmoid sinuses | 1; 2 ethmoid sinuses
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis prespecified for Efficacy 25 mm (Pivotal n=25) and all patients only. They cannot be specified per group.
Groups:
- All Patients: All Patients includes the Pilot 15 mm (n=7), Efficacy 25 mm (n=38 [Pilot n=13,Pivotal Phases n=25]) and Safety/PK 25 mm (n=5) groups.
  Pilot 15 mm and Efficacy 25 mm groups used a randomized intra-patient design wherein following FESS a non-coated splint was placed unilaterally in the ethmoid sinus opening randomized to receive the active comparator (control arm), and the drug-coated Sinexus Splint was placed contralaterally in the ethmoid sinus opening randomized to receive the intervention (treatment arm). In Pilot 15 mm group, patients in treatment arm received a 15mm length splint (220ug MF). In Efficacy 25 mm group, patients in the treatment arm received a 25mm length splint (370ug MF).
  Safety/PK group used a non-randomized design wherein following FESS a drug-coated splints (25 mm length with 370 ug MF) were placed bilaterally in both ethmoid sinus openings.
Arm/Group | All Patients
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of smoking [Count of Participants; unit: Participants]
  Never smoked | 40
  Previous smoker, stopped > 1 year ago | 5
  Current smoker | 5
Symptoms pre-op [Count of Participants; unit: Participants]
  Nasal obstruction/congestion | 40
  Discolored nasal discharge | 11
  Cough | 9
  Dental pain | 3
  Headache | 17
  Fatigue | 6
  Halitosis | 3
  Ear pain, pressure, fullness | 6
  Anosmia | 15
  Facial pain, pressure, other | 20
  Other | 22
Number of prior sinus procedures [Count of Participants; unit: Participants]
  0 | 29
  1 | 13
  2 | 7
  3 | 0
  >=4 | 1
Lund-Mackay score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay score is used to assess chronic rhinosinusitis. Each sinus (frontal, anterior ethmoidal cells, posterior ethmoidal cells, maxillary sinus, and sphenoid sinus) is scored from 0 (no abnormality), 1 (partial opacification) to 2 (complete opacification). The ostiomeatal complex is scored from 0 (not obstructed) to 2 (obstructed). Each side is graded separately. A combined score of up to 24 is possible.
  units on a scale
    Right | 6.8 (2.3)
    Left | 6.9 (2.2)
    Total | 13.6 (4.1)
Polyps [Count of Participants; unit: Participants] — Polyps at baseline is defined as either the right or left ethmoid having a polyp grade > 0
  Participants | 38

OUTCOME MEASURES:

1. Primary Outcome: Device Success Rate
Description: Device success rate defined as a ratio where the numerator is the number of successful deployments of the Sinexus Intranasal Splint and the denominator is the number of attempted sinuses. Deployment was considered successful if the implant procedure concluded with a successful splint placement on the intended side.
Time Frame: Baseline
Population: Analysis per patient.
Measure: Count of Units; unit: ethmoid sinuses
Units Other Than Participants: ethmoid sinuses
Arm/Group | Pilot 15 mm | Efficacy 25 mm | Safety/PK 25 mm
Number analyzed (Participants) | 7 | 38 | 5
Number analyzed (ethmoid sinuses) | 14 | 76 | 10
ethmoid sinuses | 14 | 76 | 10

2. Primary Outcome: Reduction in Ethmoid Sinus Inflammation
Description: Inflammation was scored by the physician using a 100-mm Visual Analog Scale (VAS) during endoscopic evaluation with range of 0 to 100mm. The term inflammation was used as a global descriptor defined to include mucosal edema, erythema, hypertrophy and polypoid changes. 0 represented no inflammation and 100mm was defined as "Severe, involving significant and extensive erythema and edema and/or hypertrophy and/or polypoid changes".
Time Frame: 21 days
Population: This measure only analyzed for Efficacy 25 mm splint (n=38). Efficacy 15 mm splint (n=7) not analyzed since it was not commercialized. Safety/PK (n=5) only evaluated for safety data.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: ethmoid sinuses
Groups:
- Efficacy (Treatment Arm, 25 mm): This group includes all ethmoid sinuses that received the 25 mm drug-coated Sinexus intranasal splint in Efficacy (Pilot Phase n=13, Pivotal Phase n=25).
- Efficacy (Control Arm, 25 mm): This group includes all ethmoid sinuses that received the 25 mm non-coated Sinexus intranasal splint in Efficacy (Pilot Phase n=13, Pivotal Phase n=25).
Arm/Group | Efficacy (Treatment Arm, 25 mm) | Efficacy (Control Arm, 25 mm)
Number analyzed (Participants) | 38 | 38
Number analyzed (ethmoid sinuses) | 38 | 38
units on a scale | 23.2 (17.7) | 35.3 (21.8)

3. Secondary Outcome: Middle Turbinate Lateralization
Description: Position of the middle turbinate was assessed using a 4-point categorical scale (medialized, normal, partially lateralized, lateralized). For Lateralized Middle Turbinate, a sinus is counted once if this occurs at least once during the 30 Day timeframe. Lateralized Middle Turbinate (worse outcome), if left unaddressed, is often the cause of sinus obstruction.
Time Frame: 30 days
Population: as for outcome 2
Measure: Count of Units; unit: ethmoid sinuses
Units Other Than Participants: ethmoid sinuses
Arm/Group | Efficacy (Treatment Arm, 25 mm) | Efficacy (Control Arm, 25 mm)
Number analyzed (Participants) | 38 | 38
Number analyzed (ethmoid sinuses) | 38 | 38
ethmoid sinuses | 2 | 6

4. Secondary Outcome: Middle Meatus Patency
Description: Patency of the middle meatus was assessed using a 3-point categorical scale (patent, narrowed, obstructed). Analysis included patent (better outcome) vs narrowed/obstructed (worse outcome).
Time Frame: 30 days
Population: as for outcome 2
Measure: Count of Units; unit: ethmoid sinuses
Units Other Than Participants: ethmoid sinuses
Arm/Group | Efficacy (Treatment Arm, 25 mm) | Efficacy (Control Arm, 25 mm)
Number analyzed (Participants) | 38 | 38
Number analyzed (ethmoid sinuses) | 38 | 38
ethmoid sinuses | 37 | 32

5. Secondary Outcome: Significant Adhesion Occurrence
Description: Adhesion formation was assessed using a 5-point categorical scale (none, small/non-obstructing, obstructing/easily separated, *dense/obstructing/difficult to separate, *severe/complete adhesion to lateral nasal wall) with "significant adhesion" denoted by *
Time Frame: 30 days
Population: as for outcome 2
Measure: Count of Units; unit: ethmoid sinuses
Units Other Than Participants: ethmoid sinuses
Arm/Group | Efficacy (Treatment Arm, 25 mm) | Efficacy (Control Arm, 25 mm)
Number analyzed (Participants) | 38 | 38
Number analyzed (ethmoid sinuses) | 38 | 38
ethmoid sinuses | 2 | 8

6. Secondary Outcome: Polypoid Tissue Changes
Description: Polyp formation in the ethmoid sinus assessed using an accepted 5-point categorical scale: 0-no visible nasal polyp (NP), 1-small amount NP confined in the middle meatus (MM); 2-multiple NP confined in MM; 3-NP extending beyond MM, within the sphenoethmoid recess not totally obstructing, or both; 4-NP completely obstructing the nasal cavity. 0 is best, and 4 is worst. When a patient's sinus has a change in polyp score at Day 30 it is counted as one.
Time Frame: 30 days
Population: as for outcome 2
Measure: Count of Units; unit: ethmoid sinuses
Units Other Than Participants: ethmoid sinuses
Arm/Group | Efficacy (Treatment Arm, 25 mm) | Efficacy (Control Arm, 25 mm)
Number analyzed (Participants) | 38 | 38
Number analyzed (ethmoid sinuses) | 38 | 38
ethmoid sinuses | 7 | 14

ADVERSE EVENTS:
Time Frame: 30 days
Description: Serious Adverse Local Tissue (SALT) response is defined as an adverse effect (bleeding, burning, or infection) occurring in the tissue of the splinted sinus cavity that is serious enough in nature or intensity as to require removal of the Sinexus intranasal splint to resolve.
Arm/Group | Pilot 15 mm | Efficacy 25 mm | Safety/PK 25 mm
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/38 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/38 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/38 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No